CLINICAL TRIAL: NCT04671004
Title: The "Concept" of Parametria: a Proposed Classification of Parametrectomy for the Treatment of Deep Infiltrating Endometriosis. A Prospective, Clinical Trial
Brief Title: The "Concept" of Parametria in the Treatment of Deep Infiltrating Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Other Study IDs: ID 3408
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Endometriosis, Parametrium, Surgery
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Deep infiltrating endometriosis (DIE) is most commonly located at the uterosacral ligaments, rectovaginal septum, pararectal space and vesicouterine fold. A nodule within the uterosacral ligaments (i.e involvement of the dorsal parametrium), increases the complexity of surgical resection. Parametrial involvement in DIE cases occurs in 25% of patients with severe endometriosis, possibly with hypogastric/sacral plexus or sciatic nerve involvement. The bladder functional impairment, after surgery for DIE involved the parametria, may vary between the 6.5% to 32.8%. Preservation of the hypogastric and pelvic splanchnic nerves represents the key aspect in pelvic surgery to prevent postoperative voiding disfunction. Several techniques for the excision of DIE have been described, but large, prospective RCTs are lacking. In particular, a clear standardization of the parametrectomy for DIE is missing. Systematic reviews on the surgical treatment of DIE demonstrated that it is impossible to compare the literature about the parametrectomy for DIE, because to unclear definitions and lack of standardization. We therefore believe it is necessary to propose a standardization of the definition of parametrectomy performed during procedures for DIE, to allow a clear comparison in the future between scientific works on surgical treatment of DIE, as already widely accepted in gynaecologic oncology with the classification of radical hysterectomy of Querleu-Morrow. In particular we believe that the parametrectomy for DIE must be described based on its anatomical extension and focused on the concepts of nerve sparing dissection, and vascular structures preservation, to reduce the risk of complications due to ischemia (i.e. ureter fistula).

Rationale A standardized description of the procedure (parametrectomy) will allow the comparison between the different techniques in terms of functionality preservation of the pelvic sympathetic and parasympathetic neural pathway. Therefore, the availability of a clear classification able to define parametria involvement during surgery would be clinically relevant, as they would allow to optimize counselling (risk of neurological consequences) and surgery planning.

Type of the study Multicentric prospective observational study. Primary objective To determinate the incidence of bladder functional impairment, after surgery for DIE involved the parametria.

Secondary objectives To classify the parametrectomy into a clear system of classification, based on anatomical landmark, and evaluate intra/postoperative complication to each classes of proposed parametrectomy.

Sample size The sample size has been calculated on the basis of the primary objective; in order to detect a proportion of bladder functional impairment of 30%, with a confidence level of 95% and a margin of error of 9%, a sample of N=100 patients is required.

Inclusion criteria - Patient scheduled for surgery for DIE

* Confirmation of DIE needed of parametrectomy at laparoscopic surgery Exclusion criteria - Patients younger than 18 years and older than 50 years at time of operation
* Refusal to answer the questionnaires
* Absence of sexual activity
* Diagnosis of multiple sclerosis
* Pre-operative urodynamic diagnosis of neurogenic bladder dysfunction Statistical analysis The sample will be described in its clinical and demographic characteristics using descriptive statistics techniques. Qualitative variables will be summarized as frequencies and percentages. Quantitative variables will be presented as mean (std.dev). Normality of data will be checked with Kolmogorov-Smirnov test. The primary objective will be achieved calculating the incidence of bladder functional impairment after surgery. The secondary objective will be achieved using descriptive statistics techniques already described.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for surgery for DIE
* Confirmation of DIE needed of parametrectomy at laparoscopic surgery

Exclusion Criteria:

* Patients younger than 18 years and older than 50 years at time of operation
* Refusal to answer the questionnaires
* Absence of sexual activity
* Diagnosis of multiple sclerosis
* Pre-operative urodynamic diagnosis of neurogenic bladder dysfunction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women scheduled for surgery for deep infiltrating endometriosis will be selected.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Bladder functional impairment | six months
  To determinate the incidence of bladder functional impairment, after surgery for DIE involved the parametria

SECONDARY OUTCOMES:
parametrectomy classification | six months
  To classify the parametrectomy into a clear system of classification, based on anatomical landmark, and evaluate intra/postoperative complication to each classes of proposed parametrectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart Rome,, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No